CLINICAL TRIAL: NCT02260518
Title: Promoting Health in Pregnancy and Postpartum Among Overweight/Obese Women
Brief Title: Promoting Health in Pregnancy and Postpartum
Acronym: HIPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Sara Wilcox, Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01HD078407 (NIH); R01HD078407 (NIH)
Record Dates: First submitted 2014-10-06; First posted 2014-10-09 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Obesity; Pregnancy; Overweight
Keywords: Gestational weight gain; Lifestyle intervention; Pregnancy; Postpartum; Physical activity; Nutrition
MeSH Terms: conditions — Obesity; Overweight; Gestational Weight Gain; Motor Activity | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle Intervention (Experimental): The intervention will focus on women gaining the recommended amount of weight, increasing physical activity to 150 minutes per week, and meeting healthy eating guidelines.
  Interventions: Behavioral: Lifestyle Intervention
- Standard Care (Other): Women in the standard care group will attend their regularly scheduled obstetric (OB) visits with their prenatal care providers and will receive monthly mailings and matched number of podcasts.
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Lifestyle Intervention — During pregnancy, participants complete one face-to-face counseling session, receive 10 behavioral podcasts, and receive weekly phone calls until delivery. Participants will be asked to attend one group session on breastfeeding. Participants will have the opportunity to participate in a private Facebook group during pregnancy and postpartum. During postpartum, participants complete one face-to-face counseling session, receive 16 behavioral podcasts, receive brief weekly check-in telephone calls for six weeks, and receive up to 8 telephone counseling calls through 6 months after delivery.
  Arms: Lifestyle Intervention
Behavioral: Standard Care — Women will receive standard nutrition counseling provided by physicians, nurses, nutritionists, and counselors from the Women, Infants, and Children (WIC) program (if applicable). They will receive a monthly study mailing that is educational in nature as well as podcasts related to a healthy pregnancy. During pregnancy, the mailings will focus on tips for a healthy pregnancy and on fetal development. During postpartum the mailings will focus on infant development and parenting. We will select a matched number of podcasts from Pea in the Podcast, commercially available podcasts. All mailings and podcasts will avoid discussion of weight, PA, or diet (except for foods to avoid in pregnancy for safety reasons).
  Arms: Standard Care

SUMMARY:
The purpose of this study is to examine the impact of a lifestyle intervention on gestational weight gain, postpartum weight loss, and other secondary outcomes relative to a usual care control group.

DETAILED DESCRIPTION:
Our study will address the following specific aims: (1) examine the impact of a lifestyle intervention on gestational weight gain and postpartum weight loss in overweight and obese women, (2) examine the impact of the intervention on physical activity (PA), dietary intake, and quality of life (QOL), (3) examine race differences in total gestational weight gain, PA, dietary intake, and QOL; and (4) examine the impact of the intervention on offspring adiposity.

ELIGIBILITY:
Inclusion Criteria:

* White or African American woman
* Overweight or obese (prepregnancy BMI: 25-45 kg/m2)
* ≤ 16 wks gestation at screening
* Age 18-44 years
* No plan to move out of the greater Columbia area in next 18 months
* Regular and consistent telephone access
* Availability for telephone calls
* Willing to accept random assignment

Exclusion Criteria:

* Uncontrolled hypertension
* Fetal anomaly
* Taking insulin for diabetes
* Uncontrolled or untreated thyroid disease
* Mental health or substance-abuse hospitalization in last 6 months
* Multiple gestation
* Persistent bleeding in the first trimester
* History of more than 3 miscarriages
* History of an eating disorder or current eating disorder
* History of an incompetent cervix
* Physical disability that prevents exercise
* Told by health care provider not to exercise
* Any other medical conditions that might be a contraindication to exercise or dietary change

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 228 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Gestational weight gain in pounds | Delivery
  Defined as delivery room weight minus pre-pregnancy weight

SECONDARY OUTCOMES:
Gestational weight gain category | Delivery
  Based on delivery room weight minus pre-pregnancy weight and categorized as Inadequate, adequate, excessive
Postpartum weight retention | Weight retained at the 6 month postpartum visit
  Defined as weight during 6 month postpartum visit minus pre-pregnancy weight
Postpartum weight retention | Weight retained at the 12 month postpartum visit
  Defined as weight during 12 month postpartum visit minus pre-pregnancy weight
Physical Activity | 32 weeks gestation
  Sense Wear Armband and self-report measure will assess physical activity
Physical Activity | 6 months postpartum
  Sense Wear Armband and self-report measure will assess physical activity
Physical Activity | 12 months postpartum
  Sense Wear Armband and self-report measure will assess physical activity
Dietary intake | 32 weeks gestation
  Two 24-hour dietary recalls using the National Cancer Institute's Automated Self-Administered 24-hour Dietary Recall (ASA-24) will assess dietary intake.
Dietary intake | 6 months postpartum
  Two 24-hour dietary recalls using the National Cancer Institute's Automated Self-Administered 24-hour Dietary Recall (ASA-24) will assess dietary intake.
Dietary intake | 12 months postpartum
  Two 24-hour dietary recalls using the National Cancer Institute's Automated Self-Administered 24-hour Dietary Recall (ASA-24) will assess dietary intake.
Depressive Symptoms | 32 weeks gestation
  Depressive symptoms will be assessed with the Edinburgh Prenatal/Postnatal Depression Scale.
Depressive Symptoms | 6 months postpartum
  Depressive symptoms will be assessed with the Edinburgh Prenatal/Postnatal Depression Scale.
Depressive Symptoms | 12 months postpartum
  Depressive symptoms will be assessed with the Edinburgh Prenatal/Postnatal Depression Scale.
Health-Related Quality of Life | 32 weeks gestation
  The Short Form-12 (SF-12) questionnaire will be used to assess quality of life.
Health-Related Quality of Life | 6 months postpartum
  The Short Form-12 (SF-12) questionnaire will be used to assess quality of life.
Health-Related Quality of Life | 12 months postpartum
  The Short Form-12 (SF-12) questionnaire will be used to assess quality of life.
Child Adiposity | 6 months postpartum
  Z-scores and skinfolds will be used to measure child adiposity.
Child Adiposity | 12 months postpartum
  Z-scores and skinfolds will be used to measure child adiposity.

OTHER OUTCOMES:
Self-efficacy for diet and physical activity | 32 weeks gestation
  Self-report measure
Self-efficacy for diet and physical activity | 6 months postpartum
  Self-report measure
Self-efficacy for diet and physical activity | 12 months postpartum
  Self-report measure
Social support for diet and physical activity | 32 weeks gestation
  Self-report measure
Social support for diet and physical activity | 6 months postpartum
  Self-report measure
Social support for diet and physical activity | 12 months postpartum
  Self-report measure
Decisional balance for diet and physical activity | 32 weeks gestation
  Self-report measure
Decisional balance for diet and physical activity | 6 months postpartum
  Self-report measure
Decisional balance for diet and physical activity | 12 months postpartum
  Self-report measure
Self-regulation for diet and physical activity | 32 weeks gestation
  Self-report measure
Self-regulation for diet and physical activity | 6 months postpartum
  Self-report measure
Self-regulation for diet and physical activity | 12 months postpartum
  Self-report measure

CONTACTS AND LOCATIONS:
Overall Officials: Sara Wilcox, PhD, Principal Investigator — University of South Carolina; Jihong Liu, Sc.D, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina Prevention Research Center, Columbia, South Carolina, United States

REFERENCES:
- [Derived] Wilcox S, Liu J, Sevoyan M, Parker-Brown J, Turner-McGrievy GM. Effects of a behavioral intervention on physical activity, diet, and health-related quality of life in postpartum women with elevated weight: results of the HIPP randomized controlled trial. BMC Pregnancy Childbirth. 2024 Dec 3;24(1):808. doi: 10.1186/s12884-024-07007-8. PMID 39627794
- [Derived] Wilcox S, Liu J, Turner-McGrievy GM, Boutte AK, Wingard E. Effects of a behavioral intervention on physical activity, diet, and health-related quality of life in pregnant women with elevated weight: results of the HIPP randomized controlled trial. Int J Behav Nutr Phys Act. 2022 Dec 9;19(1):145. doi: 10.1186/s12966-022-01387-w. PMID 36494702
- [Derived] Wilcox S, Dahl AA, Boutte AK, Liu J, Day K, Turner-McGrievy G, Wingard E. Process evaluation methods and results from the Health in Pregnancy and Postpartum (HIPP) randomized controlled trial. BMC Pregnancy Childbirth. 2022 Oct 26;22(1):794. doi: 10.1186/s12884-022-05107-x. PMID 36289464
- [Derived] Wirth MD, Liu J, Wallace MK, McLain AC, Turner-McGrievy GM, Davis JE, Ryan N, Hebert JR. Dietary Inflammatory Index and sleep quality and duration among pregnant women with overweight or obesity. Sleep. 2022 Dec 12;45(12):zsac241. doi: 10.1093/sleep/zsac241. PMID 36173829
- [Derived] Liu J, Wilcox S, Hutto B, Turner-McGrievy G, Wingard E. Effects of a lifestyle intervention on postpartum weight retention among women with elevated weight. Obesity (Silver Spring). 2022 Jul;30(7):1370-1379. doi: 10.1002/oby.23449. Epub 2022 Jun 20. PMID 35722816
- [Derived] Liu J, Wilcox S, Wingard E, Burgis J, Schneider L, Dahl A. Strategies and Challenges in Recruiting Pregnant Women with Elevated Body Mass Index for a Behavioral Lifestyle Intervention. Womens Health Rep (New Rochelle). 2020 Dec 7;1(1):556-565. doi: 10.1089/whr.2020.0089. eCollection 2020. PMID 33786522